CLINICAL TRIAL: NCT07209072
Title: Emergency Department Linkage to Care for Patients Experiencing Homelessness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, KJoseph, Principal Investigator, Denver Health and Hospital Authority
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: COMIRB 24-1764; F32HS030344 (AHRQ)
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Homelessness
Keywords: primary care; emergency department; homelessness
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Patients will receive a referral to a rapid follow up clinic at time of discharge
- Street medicine (Experimental): Patients will receive a referral to street medicine at time of discharge
  Interventions: Behavioral: Street medicine follow up

INTERVENTIONS:
Behavioral: Street medicine follow up — This intervention will use electronic health record builds to automatically send a referral to a street medicine clinic, who will attempt to contact the patient within 2 weeks.
  Arms: Street medicine

SUMMARY:
In an effort to improve access to primary care at time of discharge, patients who are homeless will be given either enhanced follow up through a street medicine team or routine follow up in clinic.

DETAILED DESCRIPTION:
Patients who experience homelessness frequently utilize the ED, but lack follow up primary care. In an effort to augment access to post-ED primary care, the investigators propose a quasi-experimental equivalent time sample study in which patients fitting certain diagnostic and inclusion criteria are allocated to either a) a referral to the Comprehensive Care Clinic at Denver Health, or b) a referral to Colorado Coalition for the Homeless (CCH) Stout Street medicine clinic. The street medicine clinic aims to lower barriers to access by locating patients on the street and providing primary care rather than asking patients to present to clinic. All patients will still receive the hospital appointment line number at time of discharge. 1 month and 3 months after index visit, the investigators will examine follow up rates at both clinics as well as secondary outcomes including ED visits, hospitalizations, and mortality through chart review of Denver Health and CCH electronic health records and CORHIO.

ELIGIBILITY:
Inclusion Criteria:

1. adult (≥18 years of age) DHMC ED patient,
2. currently unsheltered, defined as living on the streets, in a vehicle, or in another place not fit for human habitation,
3. anticipating ED discharge, with
4. a diagnosis listed below that requires short-term follow up:

   * COPD or asthma exacerbation
   * Bacterial or viral pneumonia
   * CHF with volume overload
   * SSTI
   * Dehydration requiring IV fluids
   * Hyperglycemia secondary to DM
   * Frostbite
   * First- and second-degree burns
   * Bacterial ENT infections
   * Diabetic foot infection
   * Traumatic head injury
   * Pregnancy
   * Opioid overdose
5. a stable location (i.e., an intersection, landmark, or encampment where they can be located by the street medicine team) within Denver County for at least 2 weeks.

Exclusion Criteria:

1. have altered mentation (e.g., intoxication, or secondary to medical, psychiatric, or behavioral conditions) that are unable to communicate their location, contact information, or agree to follow up.
2. are prisoners,
3. previously enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
ED visits | 1 and 3 months
  Repeat visits to the ED

SECONDARY OUTCOMES:
Inpatient hospitalizations | 1 and 3 months
  Inpatient hospitalizations at this same hospital
Mortality | 3 months
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Jason Haukoos, MD MSc, Study Director — Denver Health Medical Center
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
At this time there is no plan to share IPD. Sharing of data will be considered on a case by case basis and only de-identified data will be shared.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-10-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT07209072/Prot_SAP_ICF_001.pdf